CLINICAL TRIAL: NCT06509334
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Active-controlled Phase II Clinical Study to Evaluate the Efficacy, Safety and Tolerability of JYB1904 Injection in Adult Patients with Chronic Spontaneous Urticaria Inadequately Controlled by H1 Antihistamines
Brief Title: Trial of JYB1904 in Chronic Spontaneous Urticaria.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JYB1904-202
Record Dates: First submitted 2024-06-27; First posted 2024-07-19 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- JYB1904: Dose-1 (Experimental)
  Interventions: Drug: JYB1904
- JYB1904: Dose-2 (Experimental)
  Interventions: Drug: JYB1904
- Omalizumab (Active Comparator)
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: JYB1904 — Participants will receive JYB1904 at week0 and receive placebo at week4,8,12
  Arms: JYB1904: Dose-1
Drug: JYB1904 — Participants will receive JYB1904 at week0,8 and receive placebo at week4,12
  Arms: JYB1904: Dose-2
Drug: Omalizumab — Participants will receive Omalizumab every 4 weeks for 12 weeks
  Arms: Omalizumab

SUMMARY:
This Phase II Trial is Meant to Evaluate the Efficacy, Safety and Tolerability of JYB1904 Injection in Patients With Chronic Spontaneous Urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult subjects (≥18 years of age).
* Diagnosis of Chronic Spontaneous Urticaria(CSU) ≥ 3 months prior to Screening Visit 1 and previously inadequately controlled with a second-generation H1 antihistamine.
* Itching and hives lasting ≥ 6 weeks prior to Screening Visit 1.
* Have a UAS7 (range 0 - 42) ≥ 16, an ISS7 (range 0 - 21) ≥ 6, and an HSS7 (range 0 - 21) ≥ 6 within 7 days prior to randomization.

Exclusion Criteria:

* Induced urticaria with a defined trigger, including artificial urticaria (cutaneous scratches), cold-contact, heat-contact, solar, pressure, delayed-pressure, water-source, cholinergic, or contact urticaria
* Any other dermatological condition with chronic itching, such as atopic dermatitis, herpetic pemphigoid, herpetic dermatitis, senile itching, or psoriasis, which in the opinion of the investigator may affect the study assessment and study results
* Other conditions with symptoms of urticaria or angioedema, including but not limited to urticarial vasculitis, pigmented urticaria, erythema multiforme, mastocytosis, hereditary urticaria, or acquired/drug-induced urticaria.
* Previous allergic reaction or poor efficacy with omalizumab.
* Contraindication or hypersensitivity to antihistamines (e.g., fexofenadine, loratadine, desloratadine, cetirizine, levocetirizine, rupatadine, bilastine) or any of the ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Urticaria activity score used for 7 consecutive days(UAS7) | Baseline through 16 weeks
  Change from baseline in urticaria activity score used for 7 consecutive days (UAS7) at weeks 8, 12, and 16.Score 0-42, UAS7=0 for complete remission

SECONDARY OUTCOMES:
Urticaria activity score used for 7 consecutive days(UAS7) | Baseline through 32 weeks
  Change from baseline in UAS7 at weeks 4, 24 and 32.Score 0-42, UAS7=0 for complete remission
Itch severity score used for 7 consecutive days(ISS7) | Baseline through 32 weeks
  Change from baseline in itch severity score used for 7 consecutive days(ISS7) at weeks 4, 8, 12, 16, 24 and 32.Score 0-21, ISS7=0 for complete remission of itch
Hive severity score used for 7 consecutive days (HSS7) | Baseline through 32 weeks
  Change from baseline in hive severity score used for 7 consecutive days(HSS7) at weeks 4, 8, 12, 16, 24, 32.Score 0-21, HSS7=0 for complete remission of hives
Angioedema activity score used for 7 consecutive days(AAS7) | Baseline through 32 weeks
  Change from baseline in angioedema activity score used for 7 consecutive days(AAS7) at weeks 4, 8, 12, 16, 24, 32.Score 0-105, higher scores mean a worse outcome
Urticaria activity score used for 7 consecutive days(UAS7) | Baseline through 32 weeks
  Proportion of subjects with UAS7=0 at weeks 4, 8, 12, 16, 24, 32.Score 0-42, UAS7=0 for complete remission
Dermatology Life Quality Index(DLQI) | Baseline through 32 weeks
  Change from baseline in Dermatological Life Quality Index (DLQI) at weeks 4, 8, 12, 16, 24 and 32.Score 0-30, higher scores mean a worse outcome
Safety and tolerability | Baseline through 32 weeks
  Adverse events (AEs) and serious adverse events (SAEs)
Trends in serum total immunoglobulin E(IgE) | Baseline through 32 weeks
  Serum total IgE levels at weeks 4, 8, 12, 16, 24 and 32
Positive detection rate of anti-drug antibody (ADA) | Baseline through 32 weeks
  ADA positive detection rate at 32 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No